CLINICAL TRIAL: NCT03432039
Title: Preventing Long-term Mental Health Problems in Children Admitted With Severe Malaria at Naguru General Hospital in Uganda
Brief Title: Preventing Mental Health Problems After Childhood Severe Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC 2017-088
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation arm (Placebo Comparator): This arm will provide information about admission procedures, story telling and a follow-up phone call
  Interventions: Behavioral: Psychoeducation
- Behavioral intervention (Experimental): This arm will provide information about what invasive procedures maybe given to the child, the emotional and behavioral reactions of the child while on the ward, games and stories that the child can engage with the mother and a follow-up phone call
  Interventions: Behavioral: Behavioral

INTERVENTIONS:
Behavioral: Psychoeducation — This intervention has three phases occurring the same time as the Psychoeducation intervention. Phase I provides verbal and written information about the paediatric acute care unit services and policies. Phase II consists of: (a) verbal and written information about the general paediatric unit and its policies, and (b) a parent-child activity having ''control'' activities like reading a story not related to hospital stay. Phase III of the control program consists of a telephone call 2-3 days after discharge during which time mothers were informed that they should contact their primary healthcare providers if their children were having any problems or unusual symptoms. They also were asked to comment on their children's hospital stays during this telephone call.
  Arms: Psychoeducation arm
Behavioral: Behavioral — This is an educational-behavioural intervention that educates the parent about the children's likely emotional and behavioural problems that may result from ICU admission. Phase I will be delivered within 6 to 16 hours of admission to the hospital where caregivers are provided with information about the child's likely emotional reactions during admission in hospital. Phase II will be delivered within 2 to 16 hours of transfer to the general ward and will consist of: (a) verbal and written information to reinforce information provided in Phase I and (b) a parent-child skills building activities. Phase III of the COPE intervention program will occur 2 to 3 days after hospital discharge and will consist of a telephone call during which a 5 minute script will be read that reinforces young children's typical post-discharge emotions and behaviours and parenting behaviours which would continue to facilitate positive coping outcomes in their children.
  Arms: Behavioral intervention

SUMMARY:
This is a randomized trial in which caregivers of children suffering from malaria will be assigned to two treatment conditions to prevent mental health problems in the children. A psycho-education arm (control) and a behavioral arm (intervention). Pre- and post-intervention assessments for behavioral problems in the child and mother will be carried out.

DETAILED DESCRIPTION:
This study is designed to prevent mental health problems in children after an episode of severe malaria. The effect of the intervention on the mother's psychological wellbeing will also be assessed. Both caregivers and children will be assessed on the ward before being randomly assigned to the treatment arms. The interventions in both arms will be done in three phases with the third phase being done at home after discharge. Post-intervention assessments will be done on both the caregivers and mothers 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* aged 1.5 to 4 years
* admitted with severe malaria necessitating admission and intravenous treatment
* signed informed consent from the caregiver. Severe malaria in this study will include; cerebral malaria, severe malarial anemia, malaria with impaired consciousness (but not in coma or CM) and malaria with multiple seizures.

Exclusion Criteria:

* Living more than 50km from the hospital
* pre-existing developmental delays based on the Ten Questions Questionnaire

Ages: 18 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Presence of a behavioral problem | 6 months post-discharge
  Children whose scores on the Strength and Difficulties score for Total Problems is above 17

SECONDARY OUTCOMES:
Maternal anxiety and depression | 6 months post-discharge
  Anxiety and depression scores as measured by the Hopkins Symptom Checklist
Behavioral problems in the child | 6 months post-discharge
  Total Problems score of the Child Behavioral Checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ssenkusu JM, Hodges JS, Opoka RO, Idro R, Shapiro E, John CC, Bangirana P. Long-term Behavioral Problems in Children With Severe Malaria. Pediatrics. 2016 Nov;138(5):e20161965. doi: 10.1542/peds.2016-1965. Epub 2016 Oct 5. PMID 27940786
- [Background] Idro R, Kakooza-Mwesige A, Asea B, Ssebyala K, Bangirana P, Opoka RO, Lubowa SK, Semrud-Clikeman M, John CC, Nalugya J. Cerebral malaria is associated with long-term mental health disorders: a cross sectional survey of a long-term cohort. Malar J. 2016 Mar 31;15:184. doi: 10.1186/s12936-016-1233-6. PMID 27030124
- [Derived] Bangirana P, Birabwa A, Nyakato M, Nakitende AJ, Kroupina M, Ssenkusu JM, Nakasujja N, Musisi S, John CC, Idro R. Use of the creating opportunities for parent empowerment programme to decrease mental health problems in Ugandan children surviving severe malaria: a randomized controlled trial. Malar J. 2021 Jun 13;20(1):267. doi: 10.1186/s12936-021-03795-y. PMID 34120616